CLINICAL TRIAL: NCT06254976
Title: Correlation Between Serum Nesfatin-1 and Human Cartilage Glycoprotein-39 (YKL-40) Levels and Ultrasonographic Findings in Patients With Knee Osteoarthritis, Effect of Platelet Rich Plasma Treatment on Serum YKL-40 and Nesfatin-1 Levels
Brief Title: Serum Nesfatin-1 and Human Cartilage Glycoprotein-39 Levels in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, professor doctor, Kayseri City Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: health sciences university
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis of Knee; Degenerative Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Thirty patients were evaluated at three different time points: before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28). The assessment included the Numeric Rating Scale (NRS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), cartilage thickness measurement by ultrasonography (USG), 6-minute walk test (6MWT) parameters, and measurements of serum YKL-40 and nesfatin-1 levels.
Who Masked: Outcomes Assessor
Masking Description: The evaluations were conducted by a physical therapy and rehabilitation specialist who was blinded to the patient's treatment protocol, ensuring unbiased assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 week home exercise program (Active Comparator): Joint range of motion exercises, four-way straight leg raises, isotonic quadriceps strengthening, hamstring and quadriceps stretching exercises were given. The exercise program was demonstrated by the same physiotherapist. The patients' exercise compliance was questioned and noted.
  Interventions: Behavioral: exercise
- 2 doses of intraarticular PRP application, 1 week apart (Active Comparator): 2 doses of intra-articular 3 cc LP-PRP were applied to the patients, 1 week apart, from the inferolateral aspect of the patella, in accordance with antisepsis conditions, by a physical medicine and rehabilitation specialist.
  Interventions: Biological: intraarticular knee PRP injections

INTERVENTIONS:
Behavioral: exercise — 2 weeks of home exercise
  Arms: 2 week home exercise program
Biological: intraarticular knee PRP injections — 2 doses of intra-articular platelet rich plasma (PRP) injection, 1 week apart
  Other Names: PRP
  Arms: 2 doses of intraarticular PRP application, 1 week apart

SUMMARY:
In this study, our objective was to assess the correlation between serum human cartilage glycoprotein-39 (YKL-40) and nesfatin-1 values, the patient's clinical condition, ultrasonographic cartilage thickness measurements, and the response to PRP treatment in knee osteoarthritis (OA)

DETAILED DESCRIPTION:
The objective of this study is to assess the correlation between serum human cartilage glycoprotein-39 (YKL-40) and nesfatin-1 values, clinical condition, ultrasonographic cartilage thickness measurements, and response to PRP treatment in Knee Osteoarthritis (OA).

Thirty patients diagnosed with grade 2 and 3 knee osteoarthritis (OA) according to American College of Rheumatology (ACR) diagnostic criteria, and scheduled for leukocyte-poor platelet-rich plasma (LP-PRP) injections, were enrolled in the study. Patients were assessed at three time points: before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28). The evaluation included the Numeric Rating Scale (NRS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), cartilage thickness measurement by ultrasonography (USG), 6-minute walk test (6MWT) parameters, and measurements of serum YKL-40 and nesfatin-1 levels.

ELIGIBILITY:
Inclusion Criteria:

* Having patient consent,
* Having stage 2-3 knee osteoarthritis according to the Kellgren-Lawrence scale,
* Being diagnosed with knee osteoarthritis according to ACR (American college of Rheumatology),
* Being over the age of 18 - under the age of 75,
* Having NRS 4 and above

Exclusion Criteria:

* Those who have had knee surgery before,
* Those who have had any local injections such as physical therapy, intra-articular steroid or hyaluronic acid injection in the knee area in the last 3 months,
* Malignancies,
* Those with local infection, wound, scar in the relevant area,
* Infections, Hepatitis, Immunosuppression,
* Inflammatory arthropathies,
* Uncontrolled Hypertension, uncontrolled Diabetes Mellitus, decompensated heart failure, coronary artery disease, asthma
* Recent trauma,
* Epileptic patients,
* Pregnant women,
* Corticosteroid use,
* Avascular necrosis
* Anemia, bleeding coagulation disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum YKL-40 levels | before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28).
  It will be evaluated before and after exercise and before and after PRP. 0-14-28. day
Change in Serum nesfatin-1 levels | before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28).
  It will be evaluated before and after exercise and before and after PRP. 0-14-28. day
NRS pain score | before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28).
  Numerical Rating Scale (NRS), is basically any scale that renders a quantitative symbolization of an attribute. This type of scale is used by presenting the respondent with an ordered set from which to choose, for example, 1 to 10, coupled with anchors.The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
WOMAC score | before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28).
  It is a disease-specific measurement for knee and hip osteoarthritis. WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a personalized index with 5 questions for pain, 2 for stiffness, and 17 questions for questioning daily activities. It has different scores from 0 to 4 (0: none, 1: mild, 2: moderate, 3: severe, 4: very severe). Scale lengths of subheadings; pain=20, stiffness=8, physical function=68. Turkish validation is available . A high score indicates poor health.
6 minutes walking test | before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28).
  It is a test used to reveal submaximal functional performance. The test should be performed in a closed, quiet environment of at least 30 meters, marked every 3 meters, and in a straight corridor. The patient should be warned to wear comfortable clothes and suitable shoes. The turning points during walking should be marked with the help of a cone and the patient should be asked to go around this cone. The test is terminated by calculating the total distance walked in six minutes.A low score indicates poor health.
Cartilage thickness measurement with USG | before treatment (day 0), after exercise treatment (day 14), and after two doses of LP-PRP treatment combined with exercise treatment once a week (day 28).
  Cartilage thickness measurements (millimeter) were measured in the medial and lateral facets where the cartilage was thickest and averaged with ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Talay Çalış, Prof, Study Director — Saglik Bilimleri Universitesi; Duygu Gökbelen Bilen, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri City Hospital, Kayseri, Turkey (Türkiye)